CLINICAL TRIAL: NCT02425982
Title: Finnish Tennis Elbow Trial Pilot Study
Acronym: FINITE
Status: Completed | Type: Observational
Sponsor: University of Helsinki (Other)
Responsible Party: Principal Investigator, Tuomas Lahdeoja, MD, specialist in orthopaedics and traumatology, University of Helsinki
Other Study IDs: 65/13/03/02/2014
Record Dates: First submitted 2015-04-06; First posted 2015-04-24 (Estimated); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Tennis Elbow
Keywords: Tennis Elbow; Lateral elbow pain; Latera epicondylitis
MeSH Terms: conditions — Tennis Elbow | interventions — Conservative Treatment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Conservative treatment: Patients who will opt conservative treatment or patients treated conservatively by surgeon decision.
  Interventions: Procedure: Conservative treatment
- Operative treatment: Patients who opt for surgery when offered.
  Interventions: Procedure: Operative treatment

INTERVENTIONS:
Procedure: Operative treatment — The exact treatment depends on the surgeon, but the majority are anticipated to be elbow arthroscopy followed by either arthroscopic or open extensor carpi radialis brevis release.
  Groups: Operative treatment
Procedure: Conservative treatment — The treatment consists of physiotherapy, activity modification, pain medication and watchful waiting. Injection therapies will be avoided.
  Groups: Conservative treatment

SUMMARY:
The study aims to investigate the natural course and the results of operative treatment of chronic tennis elbow (TE). Chronic is defined as symptoms having lasted for more than a year. The investigators will also study the effect of pain catastrophising on the subjective outcome, the patient acceptable symptomatic state and the response shift phenomenon in TE. The study will also ascertain the feasibility of a multi-center randomised, controlled trial (RCT), and test and refine the co-operation and interaction of the planned RCT centers.

DETAILED DESCRIPTION:
Objectives:

1. To study the natural course of tennis elbow/spontaneous recovery of chronic (lasting for over 12 months) tennis elbow and the results of surgery in a pragmatic setting.
2. To investigate the patients' expectations of the treatment, and define the patient acceptable symptomatic state, or PASS, in tennis elbow.
3. To investigate the effect of pain behaviour on treatment results and PASS.
4. To delineate the existence of a potential "response shift" -phenomenon in patients with a tennis elbow.
5. To determine the feasibility of a prospective, placebo-controlled, randomised trial by finding out the actual number of patients in each center and those that may be suitable for the FINITE-RCT. The investigators will also test the functioning and response of the planned outcome measures in this environment and for this purpose.

Study setting The study is carried out as a prospective open-label multi-center cohort study.

The study was originally planned with a follow-up up to 10 years, but the cost-benefit of the long term follow-up was evaluated after the completion of one year data collection, and the decision was made to shorten the follow-up to include two year data, but no further follow-ups.

ELIGIBILITY:
Inclusion Criteria:

1. Clinically diagnosed tennis elbow defined as: Pain on the lateral side of the elbow, made worse by pressure applied on the lateral epicondyle of the humerus and during resisted extension of the wrist or when making a fist with the elbow joint straight.
2. Duration of symptoms over 10 months
3. Age between 35 and 60 years
4. Ability to fill in Finnish questionnaires
5. Written informed consent

Exclusion Criteria:

1. Earlier fracture or dislocation in the elbow joint area
2. Earlier surgical treatment of the same elbow joint
3. Congenital deformity in the elbow
4. Systemic muscle, tendon, nerve or joint disease
5. Other problems causing pain the elbow joint:

   1. Pain in the medial epicondyle of the elbow
   2. Pain in the biceps muscle tendon
   3. Painful snapping or crepitus of elbow joint
   4. Instability of elbow joint (table top, posterolateral drawer test)
6. A passive movement limitation of more than 10 degrees in the elbow joint
7. Abnormal finding in an elbow joint X-ray. An elbow joint X-ray is a routine examination of elbow symptoms.

Ages: 35 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: All patients who seek advice or treatment at the outpatient clinics of the centers taking part in the study will be assessed for eligibility. Those fulfilling the criteria defined below will be asked to participate.
Sampling Method: Non-Probability Sample
Enrollment: 99 (Actual)
Dates: Start 2015-08; Primary Completion 2018-03-15 (Actual); Study Completion 2018-03-15 (Actual)

PRIMARY OUTCOMES:
Global improvement | 6 months
  A six-point Likert scale (much worse - worse - no change - better - much better - complete recovery) will be used and the patient is asked how the elbow symptoms are compared to the situation at the time of the initial visit and inclusion to the study.
Oxford Elbow Score | 6 months
  Oxford Elbow Score (OES) is a three-dimensional questionnaire consisting of 12 multiple-choice questions answered by the patient. OES has been validated for patients with surgically treated elbow problems. OES is the most robust elbow-specific PROM available currently.

SECONDARY OUTCOMES:
QuickDASH | up to 2 years
  QuickDASH is a validated patient reported outcome measure of the function the upper extremities. It consists of 11 questions and 4 work-related questions. An approved Finnish translation has been made earlier. The outcome measure will be assessed as a secondary outcome at 6, 12, 26 and 52 weeks and then at 2, 3, 4, 5 and 10 years.
Success rate | up to 2 years
  Success is defined at any follow-up time point as patients who report "much better" or "complete recovery" in the second primary outcome question.
Relapses | up to 2 years
  Relapses are calculated from the Likert answers so that if the patient reports "much better" or "completely healed" at time point X and the answer is "better" or any of the poorer alternatives on follow-up point X+1, this is interpreted as a relapse for X+1 point in time. Relapses are calculated for each follow-up point in time and the patients are considered to remain in "relapse" until they report "much better" or "completely healed".
Satisfaction with the treatment process | up to 2 years
  this is evaluated with the question "On a scale of 0 to 10, (with 10 on as 'very satisfied' and 0 as 'very dissatisfied'), how satisfied are you with the treatment you have received as a whole?" The outcome measure will be assessed as a secondary outcome at 6, 12, 26 and 52 weeks and then at 2, 3, 4, 5 and 10 years
Time off work | up to 2 years
  Number of sick leave days due to elbow symptoms.
Complications and adverse effects | up to 2 years
  Complications and adverse events related to treatment of the elbow. Predefined complications are: infection, iatrogenic injuries (especially nerve), crps, anaesthetic complications.
Global improvement | up to 2 years
  A six-point Likert scale (much worse - worse - no change - better - much better - complete recovery) will be used and the patient is asked how the elbow symptoms are compared to the situation at the time of the initial visit and inclusion to the study. The outcome measure will be assessed at 6, 12, 26 and 52 weeks and then at 2, 3, 4, 5 and 10 years
Oxford Elbow Score | up to 2 years
  OES will be assessed as a secondary outcome at 6, 12, 26 and 52 weeks and then at 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Teppo LN Järvinen, MD, professor, Study Director — Helsinki University, Helsinki University Central Hospital; Tuomas Lähdeoja, MD, Principal Investigator — Helsinki University, Helsinki University Central Hospital; Mikko Salmela, MD, Principal Investigator — Helsinki University, Helsinki University Central Hospital; Teemu Karjalainen, MD, PhD, Principal Investigator — Central Finland Central Hospital; Pirjo Toivonen, coordinator, Principal Investigator — Helsinki University, Hatanpää Hospital
Locations (12):
- Finland (12):
  - Töölö Hospital, Helsinki, Uusimaa
  - North Karelia Central Hospital, Joensuu
  - Central Finland Central Hospital, Jyväskylä
  - Kymenlaakso Central Hospital, Kotka
  - Kuopio Unversity Hospital, Kuopio
  - Päijät-Häme Central Hospital, Lahti
  - Oulu University Hospital, Oulu
  - Satakunta Central Hospital, Pori
  - Seinäjoki Central Hospital, Seinäjoki
  - Hatanpää Hospital, Tampere
  - Tampere Unversity Hospital, Tampere
  - Turku University Hospital, Turku

REFERENCES:
- [Derived] Karjalainen T, Lahdeoja T, Salmela M, Ardern CL, Juurakko J, Jarvinen TL, Taimela S; FINITE investigators. Minimal important difference, patient acceptable symptom state and longitudinal validity of oxford elbow score and the quickDASH in patients with tennis elbow. BMC Med Res Methodol. 2023 Jul 6;23(1):158. doi: 10.1186/s12874-023-01934-4. PMID 37415100